CLINICAL TRIAL: NCT03520257
Title: A Randomized Clinical Study of Apatinib Plus Radiotherapy vs. Apatinib in the Treatment of Hepatocellular Carcinoma With BCLC-C Stage I and Stage II Portal Vein Tumor Thrombus
Brief Title: The Study of Apatinib Plus Radiotherapy vs. Apatinib in the Treatment of Hepatocellular Carcinoma With BCLC-C Stage I and Stage II Portal Vein Tumor Thrombus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, TaoBai, Researcher, Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GuangxiMU-HCC
Record Dates: First submitted 2018-04-17; First posted 2018-05-09 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — apatinib; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apatinib Plus Radiotherapy (Experimental)
  Interventions: Drug: Apatinib; Device: Radiotherapy
- Apatinib (Other)
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Apatinib, a small molecule anti-angiogenic targeted drug that has been demonstrated to be safe and effective after failure of standard chemotherapy for advanced gastric cancer, has been initially successful in phase II clinical trials for the treatment of unresectable advanced HCC patients. The efficacy of ralfiny in the treatment of Oriental population (ORIENTAL study) is better. The randomized, double-blind, multi-center phase III clinical study of apatinib second-line treatment of advanced hepatocellular carcinoma showed a good efficacy and safety. Currently, Phase III clinical studies of apatinib in HCC patients undergoing systemic chemotherapy or sorafenib treatment have progressed. Initial results also showed good efficacy and safety.
Device: Radiotherapy — Radiotherapy of tumors and portal vein tumor thrombi can promote further tumor shrinkage, and at the same time, the physiological basis for the recanalization of the original tumor thrombus itself will result in necrosis and fibrosis of the tumor thrombus, completely blocking the blood supply to the tumor portal vein. As a result, blood supply to the other side of the portal vein increases, and hepatocyte regeneration in a healthy liver is promoted, so that the patient can obtain surgical opportunities.
  Arms: Apatinib Plus Radiotherapy

SUMMARY:
This study uses to suppress the growth of tumors, extend the patient's survival time and improve the quality of life as much as possible. Through the treatment, the patient is given the chance to undergo surgical resection, thereby more effectively prolonging the OS. Apatinib is a small-molecule VEGFR tyrosine kinase inhibitor. It mainly treats malignant tumors by inhibiting VEGFR and exerting anti-angiogenic effects. Preclinical studies have shown that its anti-tumor effect is better than that of the similar drug PTK787. Phase II studies of hepatocellular carcinoma have initially demonstrated the effectiveness and safety of apatinib in the treatment of advanced HCC. Radiotherapy of tumors and portal vein tumor thrombi can promote further tumor shrinkage, and at the same time, the physiological basis for the recanalization of the original tumor thrombus itself will result in necrosis and fibrosis of the tumor thrombus, completely blocking the blood supply to the tumor portal vein. As a result, blood supply to the other side of the portal vein increases, and hepatocyte regeneration in a healthy liver is promoted, so that the patient can obtain surgical opportunities. Based on the therapeutic potential of apatinib and radiotherapy, we designed a prospective exploratory clinical study of this patient with advanced liver cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years old;
2. An unresectable HCC patient who is in strict compliance with the criteria for diagnosis and treatment of primary liver cancer (2011 edition) or who has been diagnosed by pathological or cytological examination and has at least one measurable lesion;
3. Child-Pugh Liver Function Rating: Grade A or better Grade B (≤ 7 points);
4. Cheng's type I and type II (imaging evaluation of the tumor portal vein tumors did not reach the contralateral portal vein branch, and embolization does not exceed 50% of the portal vein diameter) PVTT BCLC-C patients;
5. Clinical evaluation cannot tolerate radical surgical resection;
6. The tumor is confined to the hepatic liver;
7. The first patient who had not received any anti-cancer comprehensive treatment before;
8. ECOG PS score: 0-1 points;
9. The expected survival period is ≥ 3 months;
10. The normal function of the major organs is the following:

    * Blood tests:

      1. HGB≥90 g/L;
      2. Neutrophil absolute count (ANC) ≥ 1.5 × 109/L;
      3. PLT≥60×109/L;
    * Biochemical tests:

      1. ALB ≥ 29 g/L;
      2. ALT and AST <2.5ULN;
      3. TBIL ≤ 2ULN;
      4. Creatinine ≤1.5ULN; (Child-Pugh can only have 2 points for both albumin and bilirubin)
11. Subjects voluntarily joined the study and signed informed consent. Good compliance and follow-up.

Exclusion Criteria:

1. Pregnancy or breast-feeding women, or those who are unwilling or unable to take effective contraceptive measures if they have fertility, women who are of child-bearing age will have a pregnancy test (+) within 7 days before enrollment;
2. Participated in other drug clinical trials within 8 weeks before the start of the study;
3. History of other malignancies in the past 5 years;
4. Ascites with clinical symptoms, which require therapeutic paracentesis or drainage;
5. People with high blood pressure who are unable to fall within the normal range after treatment with antihypertensive drugs (systolic blood pressure>140 mmHg, diastolic blood pressure>90 mmHg);
6. Arrhythmia with grade II or higher myocardial ischemia or myocardial infarction and poor control;
7. In accordance with NYHA criteria III-IV heart failure or cardiac ultrasound examination: LVEF (left ventricular ejection fraction) <50%;
8. No other serious heart, lung, brain, kidney dysfunction;
9. Has a variety of factors that affect oral medications (eg, inability to swallow, chronic diarrhea, and intestinal obstruction, which significantly affect drug use and absorption);
10. In the past 6 months, there was a history of digestive tract bleeding or a clear tendency to gastrointestinal bleeding. For example, esophageal varices, local active ulcer lesions, fecal occult blood ≥ (++) with risk of bleeding may not be included in the group; If fecal occult blood (+) requires gastroscopy;
11. Incidental arterial/venous thromboembolic events such as cerebrovascular accidents (including transient ischemic attacks), deep venous thrombosis, and pulmonary embolism within the first 6 months of study initiation;
12. Coagulation abnormalities (INR> 1.5 or prothrombin time (PT)> ULN + 4 seconds) with bleeding tendency or receiving thrombolytic or anticoagulant therapy;
13. Urinary cues suggest that urinary protein ≥ ++ and confirm 24-hour urinary protein quantification> 1.0 g;
14. Those who have a history of abuse of psychotropic substances and are unable to get rid of or have a history of mental disorders;
15. Existence of immune diseases or HIV infection;
16. The investigator judges other situations that may affect the conduct of clinical studies and the findings of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5 years

IPD SHARING:
Plan to Share IPD: Undecided